CLINICAL TRIAL: NCT00365274
Title: A Phase II Study of SGN-30 in Combination With CHOP in Anaplastic Large Cell Lymphoma
Brief Title: SGN-30 and Combination Chemotherapy in Treating Patients With Newly Diagnosed Anaplastic Large Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00162; 2005-0627 (Other: UT MD Anderson Cancer Center); N01CM62202 (NIH); N01CM17003 (NIH)
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2013-11

CONDITIONS: Anaplastic Large Cell Lymphoma
Keywords: non-Hodgkin's lymphoma; NHL; murine monoclonal antibody; mAb; SGN-30; CHOP; Cyclophosphamide; Doxorubicin Hydrochloride; Vincristine; Prednisone; anaplastic large cell lymphoma; Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Anaplastic; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, B-Cell; Lymphoma, T-Cell; Antibodies; Antibodies, Monoclonal; Immunologic Factors; Physiological Effects of Drugs; Pharmacologic Actions; Immunosuppressive Agents; Antirheumatic Agents; Therapeutic Uses; Antineoplastic Agents, Alkylating; Alkylating Agents; Molecular Mechanisms of Pharmacological Action; Antineoplastic Agents; Myeloablative Agonists; Antibiotics; Antineoplastic
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, Large B-Cell, Diffuse; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, B-Cell; Lymphoma, T-Cell | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SGN-30 + Combination Chemotherapy (Experimental): Monoclonal antibody SGN-30 monotherapy: SGN-30 12 mg/kg weekly intravenously(IV) over 2 hours once weekly for 3 weeks.
  SGN-30 and CHOP chemotherapy: Beginning 1 week after completion of monoclonal antibody SGN-30 monotherapy, SGN-30 12 mg/kg IV over 2 hours on day 1 and CHOP chemotherapy comprising cyclophosphamide IV over 1 hour, doxorubicin hydrochloride IV over 15 minutes, and vincristine IV over 15 minutes on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for 6-8 courses.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin hydrochloride; Drug: vincristine sulfate; Drug: prednisone; Drug: SGN-30

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV 750 mg/m^2 day 1
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: Doxorubicin hydrochloride — Given 50 mg/m^2 IV day 1
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: vincristine sulfate — Given 1.4 mg/m^2 IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: prednisone — 100 mg orally daily days 1 - 5
  Other Names: DeCortin; Deltra
Drug: SGN-30 — 12 mg/kg weekly IV over 2 hours once weekly for 3 weeks.
  Other Names: Monoclonal antibody SGN-30 monotherapy

SUMMARY:
This phase II trial is studying how well giving SGN-30 together with combination chemotherapy works in treating patients with newly diagnosed anaplastic large cell lymphoma. Monoclonal antibodies, such as SGN-30, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving SGN-30 together with combination chemotherapy may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of monoclonal antibody SGN-30 in combination with cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone (CHOP) in patients with newly diagnosed anaplastic large cell lymphoma (ALCL).

II. Determine the safety of combining monoclonal antibody SGN-30 with CHOP chemotherapy.

SECONDARY OBJECTIVES:

I. Determine whether monoclonal antibody SGN-30 can induce apoptosis of ALCL cells in vivo.

II. Determine the response duration in patients treated with this regimen.

III. Correlate response with pretreatment serum CD30 levels.

IV. Determine response to single-agent monoclonal antibody SGN-30.

OUTLINE: This is a multicenter study. Patients are stratified according to anaplastic large cell kinase (ALK) status (positive vs negative).

Monoclonal antibody SGN-30 monotherapy: Patients receive monoclonal antibody SGN-30 IV over 2 hours once weekly for 3 weeks.

Monoclonal antibody SGN-30 and CHOP chemotherapy: Beginning 1 week after completion of monoclonal antibody SGN-30 monotherapy, patients receive monoclonal antibody SGN-30 IV over 2 hours on day 1 and CHOP chemotherapy comprising cyclophosphamide IV over 1 hour, doxorubicin hydrochloride IV over 15 minutes, and vincristine IV over 15 minutes on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for 6-8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed systemic anaplastic large cell lymphoma (ALCL)
* Tissue available for the determination of anaplastic large cell kinase (ALK) status [t(2;5), ALK-NPM translocation] prior to study entry
* Prior steroids or topical treatments are allowed. Patients who are on chronic steroid therapy may receive concomitant steroids provided they have been on a stable dosage for at least 3 months prior to enrollment
* Measurable disease, defined as >= 1 lesion that can be accurately measured in >= 1 dimension (longest diameter to be recorded) as >= 20 mm by conventional techniques or as >= 10 mm by spiral CT scan
* The Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1 OR Karnofsky PS 70-100%
* White Blood Count (WBC) >= 3,000/mm³
* Absolute neutrophil count >= 1,500/mm³
* Platelet count >= 100,000/mm³ (unless due to lymphoma [i.e., splenomegaly and/or bone marrow involvement])
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* AST or ALT =< 2.5 times ULN
* Creatinine =< 1.5 times ULN (unless due to lymphoma) OR creatinine clearance >=60 mL/min
* Left ventricular ejection fraction (LVEF) >= 50%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment

Exclusion Criteria:

* No rapidly progressing disease or bulky disease, defined as a mass of > 7 cm in largest diameter
* No primary cutaneous ALCL
* No known brain metastases
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to monoclonal antibody SGN-30
* No uncontrolled intercurrent illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would preclude study compliance
* No prior or other concurrent malignancy with < 90% probability of survival at 5 years
* No other concurrent anticancer agents or therapies
* No prior chemotherapy for ALCL
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Fanale, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 9, 2006 to February 26, 2009. All recruitment was done in medical clinics.
Pre-assignment Details: The six participants were registered at UT MD Anderson Cancer Center prior to early study termination although recruitment was open to multi-centers.
Groups:
- SGN-30 + Combination Chemotherapy: Monoclonal antibody SGN-30 monotherapy: SGN-30 12 mg/kg weekly intravenously (IV) over 2 hours once weekly for 3 weeks.
  SGN-30 and CHOP chemotherapy: Beginning 1 week after completion of monoclonal antibody SGN-30 monotherapy, SGN-30 12 mg/kg IV over 2 hours on day 1 and CHOP chemotherapy comprising cyclophosphamide IV over 1 hour, doxorubicin hydrochloride IV over 15 minutes, and vincristine IV over 15 minutes on day 1 and oral prednisone once daily on days 1-5. Treatment repeats every 21 days for 6-8 courses.
Period: Overall Study
Arm/Group | SGN-30 + Combination Chemotherapy
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SGN-30 + Combination Chemotherapy
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 36 [20 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) defined as the proportion of participants experiencing a Complete Response (CR) or Partial Response to a regimen of SGN-3- + CHOP using International Workshop Response Criteria (IWG) for Non-Hodgkin's Lymphomas (NHL). The IWG criteria (Cheson et al 2007) for a CR is a complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. A PR is at least a 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses, no increase should be observed in the size of other nodes, liver or spleen, and no new sites of disease should be observed.
Time Frame: Up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | SGN-30 + Combination Chemotherapy
Number analyzed (Participants) | 6
percentage of participants
  Complete Response | 83
  Partial Response | 17

ADVERSE EVENTS:
Time Frame: 2 years and 11 months
Arm/Group | SGN-30 + Combination Chemotherapy
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SGN-30 + Combination Chemotherapy (N=6)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Elevated ALT, SGPT (Blood and lymphatic system disorders) | 1 — alanine aminotransferase (ALT) or serum glutamic-pyruvic transaminase (SGPT)
Elevated Bilirubin (Blood and lymphatic system disorders) | 1
Blurred Vision (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Edema: head and neck (Investigations) | 1
Fatigue (General disorders) | 3
Fever without neutropenia (Infections and infestations) | 2
Elevated Hemoglobin (Blood and lymphatic system disorders) | 1
Hot flashes (Reproductive system and breast disorders) | 1
Hyperglycemia (Blood and lymphatic system disorders) | 2
Hypoglycemia (Blood and lymphatic system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Elevated Leukocytes (Blood and lymphatic system disorders) | 3
Memory impairment (Psychiatric disorders) | 2
Mood alteration (depression) (Psychiatric disorders) | 1
Mucositis, oral cavity (Respiratory, thoracic and mediastinal disorders) | 4
Nausea (Gastrointestinal disorders) | 2
Neuropathy: motor (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 2
Elevated Neutrophils (ANC/AGC) (Blood and lymphatic system disorders) | 2 — Absolute neutrophil count (ANC)/Absolute Granulocyte Count (AGC)
Ocular/visual (other) (Eye disorders) | 1
Pain (Musculoskeletal and connective tissue disorders) | 4 — Back, Bone, Face, Head, Muscle, and Other
Elevated Platelets (Blood and lymphatic system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Rigors/chills (Investigations) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Watery Eye (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less